CLINICAL TRIAL: NCT00462761
Title: Phase I Open-Label, Sequential Dose Escalation Study Investigating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AC220 When Administered Daily to Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: A Phase I Study of AC220 in Patients With Relapsed/Refractory Acute Myeloid Leukemia Regardless of FLT3 Status
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0001
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia; Leukemia; Myelodysplastic Syndrome; AML; MDS
Keywords: RTK; kinase; inhibitor; tyrosine; acute; FLT3; AC220; pharmacokinetic; pharmacokinetics; PK; pharmacodynamic; pharmacodynamics; mutations; PD; receptor; class III; relapsed; refractory; t(8;21); q22;q22; AML1/ETO; t(16;16; p13;q22; CBFbeta/MYH11; inv(16); p13q22; 11q23; dysplasia; myeloid; myelomonocytic; monoblastic; monocytic; erythroid; erythroleukemia; megakaryoblastic; basophilic; panmyelosis; myelofibrosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Myelodysplastic Syndromes; Recurrence; Aortic aneurysm, familial thoracic 4; Leukemia, Erythroblastic, Acute; Primary Myelofibrosis | interventions — quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AC220 (Experimental): Determine safety, tolerability and pharmacokinetic (PK) parameters of AC220
  Interventions: Drug: AC220

INTERVENTIONS:
Drug: AC220 — Powder in bottle formulation supplied as 50mg or 350 mg in glass, crimped serum vials. Requires reconstitution by a pharmacist, and must be stored securely and protected from light.
  Other Names: Quizartinib

SUMMARY:
Patients received oral AC220 daily for 14 days to study the side effects, tolerability and best dose for treating relapsed or refractory acute myeloid leukemia, regardless of FLT3 status.

DETAILED DESCRIPTION:
This is a multi-center clinical study conducted in the USA and two international sites. This open-label, dose escalation study was designed to characterize the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of orally administered AC220 as a single agent given daily for 14 days. Cohorts of 3 patients received AC220 until dose limiting toxicity was noted (DLT). At that point cohorts expanded to 6 patients until MTD was determined. Patients not experiencing DLT or significant disease progression at Day 15 may have continued receiving AC220 at the discretion of the Investigator and Sponsor. FLT3 positive and negative patients were allowed to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age ≥ 18 years;
2. Histopathologically documented primary or secondary AML, as defined by WHO criteria (Jaffe et al, 2001), confirmed by pathology review at treating institution, meeting at least one of the following:

   1. Refractory to at least 1 cycle of induction chemotherapy, or
   2. Relapsed after at least 1 cycle of induction chemotherapy, or
   3. Patient is not, according to the clinical judgment of the Principal Investigator, a candidate for induction chemotherapy due to age, comorbidity, or other factors;
3. Patients for whom no standard therapies are anticipated to result in a durable remission, or who have failed potentially curative therapy, or who refuse standard therapy or patients for whom there is no known therapy of documented treatment benefit;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-3;
5. In the absence of rapidly progressing disease, the interval from prior treatment to time of AC220 administration should be at least 2 weeks for cytotoxic agents (other than hydroxyurea, per Section 8.8), or at least 5 half-lives for noncytotoxic agents;
6. Persistent chronic clinically significant toxicities from prior chemotherapy or surgery must be less than Grade 2;
7. Serum creatinine ≤ 2.0 mg/dL;
8. Total serum bilirubin ≤ 1.5 × ULN unless considered due to Gilbert's syndrome or leukemic organ involvement;
9. Serum AST or ALT ≤ 3.0 × ULN unless considered due to leukemic organ involvement;
10. Females of childbearing potential must have a negative pregnancy test (urine β-hCG);
11. Females of childbearing potential and sexually mature males must agree to use a medically accepted method of contraception throughout the study;
12. Written informed consent must be provided.

Exclusion Criteria:

1. Histologic diagnosis of acute promyelocytic leukemia;
2. Clinically active central nervous system leukemia;
3. Persistent clinically significant toxicity from prior chemotherapy that is Grade 2 or higher by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v3);
4. Bone marrow transplant within 2 months prior to study;
5. Active, uncontrolled infection;
6. Major surgery within 4 weeks prior to study;
7. Radiation therapy within 4 weeks prior to, or concurrent with, study;
8. Human immunodeficiency virus positivity;
9. Active hepatitis B or C or other active liver disease;
10. Women who are pregnant, lactating, or unwilling to use contraception if of childbearing potential;
11. Medical condition, serious intercurrent illness, or other extenuating circumstance that, in the judgment of the Principal Investigator, could jeopardize patient safety or interfere with the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Daiichi Sankyo
Locations (5):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Nebraska Medical Center, Omaha, Nebraska
  - MD Anderson Cancer Center, Houston, Texas
- Georgia (2):
  - Chemotherapy and Immunotherapy Clinic, Tbilisi
  - Hematology and Chemotherapy Clinic, Tbilisi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Cortes JE, Kantarjian H, Foran JM, Ghirdaladze D, Zodelava M, Borthakur G, Gammon G, Trone D, Armstrong RC, James J, Levis M. Phase I study of quizartinib administered daily to patients with relapsed or refractory acute myeloid leukemia irrespective of FMS-like tyrosine kinase 3-internal tandem duplication status. J Clin Oncol. 2013 Oct 10;31(29):3681-7. doi: 10.1200/JCO.2013.48.8783. Epub 2013 Sep 3. PMID 24002496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 76 participants who met all inclusion and no exclusion criteria were enrolled and treated in the study at 4 clinical sites in the United States and 2 sites in the Republic of Georgia.
Groups:
- Quizartinib: Participants initially received quizartinib (AC220) on an intermittent dosing (ID) schedule (14 days on treatment followed by 14 days off treatment) up to a maximum of 200 mg/day.
  Following a protocol amendment, participants then received a starting dose of 300 mg/day quizartinib on an ID regimen or received a starting dose of 200 mg/day quizartinib for 28 days (1 cycle) on a continuous dosing schedule.
Period: Overall Study
Arm/Group | Quizartinib
Started | 76
Completed | 0
Not Completed | 76
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 9
Not completed — Physician Decision | 5
Not completed — Disease progression | 43
Not completed — Death | 12
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Quizartinib
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (17.1)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  18 to 60 years | 39
  61 to 75 years | 31
  >75 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 68
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Treatment Related Adverse Events Following Oral Administration of Quizartinib in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Time Frame: Baseline up to 30 days post last dose
Population: Safety events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib
Number analyzed (Participants) | 76
Participants
  At Least 1 Treatment-Related Adverse Event | 39
  General disorders & administration site conditions | 11
  Pyrexia | 2
  Fatigue | 4
  Oedema peripheral | 6
  Asthenia | 1
  Chills | 1
  Malaise | 1
  Gastrointestinal disorders | 21
  Nausea | 12
  Diarrhoea | 6
  Vomiting | 8
  Abdominal pain | 3
  Abdominal pain upper | 2
  Dyspepsia | 3
  Constipation | 1
  Abdominal distension | 2
  Gastrointestinal haemorrhage | 1
  Gastrooesophageal reflux disease | 1
  Abdominal discomfort | 1
  Oral mucosal blistering | 1
  Epigastric discomfort | 1
  Retching | 1
  Respiratory, Thoracic, and Mediastinal Disorders | 2
  Haemoptysis | 1
  Dyspnoea exertional | 1
  Blood and Lymphatic System Disorders | 4
  Anaemia | 3
  Thrombocytopenia | 1
  Pancytopenia | 1
  Skin and Subcutaneous Tissue Disorders | 8
  Periorbital odema | 1
  Swelling face | 1
  Alopecia | 2
  Dry skin | 1
  Increased tendency to bruise | 1
  Hair colour changes | 1
  Hidradenitis | 1
  Photosensitivity reaction | 1
  Infections and Infestations | 1
  Pneumonia | 1
  Lung infection | 1
  Metabolism and Nutrition Disorders | 7
  Hypokalaemia | 2
  Anorexia | 5
  Hyperglycaemia | 1
  Hypoalbuminaemia | 1
  Nervous System Disorders | 12
  Headache | 2
  Dizziness | 1
  Dysgeusia | 8
  Hypoaesthesia | 1
  Neuropathy peripheral | 1
  Dysarthria | 1
  Investigations | 11
  Electrocardiogram QT prolonged | 9
  Blood bilirubin increased | 1
  Hepatic enzyme increased | 1
  Psychiatric Disorders | 1
  Insomnia | 1
  Cardiac Disorders | 1
  Right ventricular dysfunction | 1
  Injury, Poisoning, and Procedural Complications | 1
  Contusion | 1
  Eye Disorders | 1
  Eyelid oedema | 1
  Hepatobiliary Disorders | 3
  Hyperbilirubinaemia | 3
  Jaundice | 1

2. Primary Outcome: Number of Participants With Treatment-emergent Treatment-related Grade 3 or 4 Adverse Events By At Least 10% of All Participants By Dose Group Following Oral Administration of Quizartinib in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Time Frame: Baseline up to 30 days post last dose
Population: Safety events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Quizartinib 12-135 mg ID: Participants received quizartinib (AC220) with doses ranging from 12-135 mg on an intermittent dosing (ID) schedule.
- Quizartinib 200-450 mg ID: Participants received quizartinib (AC220) with doses ranging from 200-450 mg on an intermittent dosing (ID) schedule.
- Quizartinib 200-300 mg CD: Participants received quizartinib (AC220) with doses ranging from 200-300 mg on a continuous dosing (CD) schedule.
- Total: All participants who received quizartinib, regardless of dosage or dosing schedule.
Arm/Group | Quizartinib 12-135 mg ID | Quizartinib 200-450 mg ID | Quizartinib 200-300 mg CD | Total
Number analyzed (Participants) | 35 | 16 | 25 | 76
Participants
  Nausea : All Grades | 6 | 3 | 3 | 12
  Nausea : Grade 3-4 | 0 | 0 | 0 | 0
  Electrocardiogram QT prolonged : All Grades | 1 | 0 | 8 | 9
  Electrocardiogram QT prolonged : Grade 3-4 | 0 | 0 | 4 | 4
  Dysgeusia : All Grades | 4 | 1 | 3 | 8
  Dysgeusia : Grade 3-4 | 0 | 0 | 0 | 0
  Vomiting : All Grades | 3 | 3 | 2 | 8
  Vomiting : Grade 3-4 | 1 | 0 | 0 | 1
  Anorexia : All Grades | 3 | 1 | 1 | 5
  Anorexia : Grade 3-4 | 1 | 0 | 0 | 1
  Fatigue : All Grades | 2 | 1 | 1 | 4
  Fatigue : Grade 3-4 | 1 | 0 | 1 | 2
  Anaemia : All Grades | 2 | 1 | 0 | 3
  Anaemia : Grade 3-4 | 2 | 1 | 0 | 3
  Hypokalaemia : All Grades | 2 | 0 | 0 | 2
  Hypokalaemia : Grade 3-4 | 1 | 0 | 0 | 1
  Pyrexia : All Grades | 2 | 0 | 0 | 2
  Pyrexia : Grade 3-4 | 1 | 0 | 0 | 1
  Eyelid oedema : All Grades | 0 | 1 | 0 | 1
  Eyelid oedema : Grade 3-4 | 0 | 1 | 0 | 1
  Hypoalbuminaemia : All Grades | 0 | 1 | 0 | 1
  Hypoalbuminaemia : Grade 3-4 | 0 | 1 | 0 | 1
  Lung infection : All Grades | 0 | 1 | 0 | 1
  Lung infection : Grade 3-4 | 0 | 1 | 0 | 1
  Pancytopenia : All Grades | 1 | 0 | 0 | 1
  Pancytopenia : Grade 3-4 | 1 | 0 | 0 | 1
  Photosensitivity reaction : All Grades | 0 | 0 | 1 | 1
  Photosensitivity reaction : Grade 3-4 | 0 | 0 | 1 | 1
  Thrombocytopenia : All Grades | 0 | 0 | 1 | 1
  Thrombocytopenia : Grade 3-4 | 0 | 0 | 1 | 1

3. Secondary Outcome: Number of Participants Achieving a Best Disease Response by Dose Cohort in Terms of Progressive Disease Following Oral Administration of Quizartinib in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Progressive disease response criteria included doubling of blast count % in bone marrow (biopsy or aspirate) from baseline; considering measurements starting on Study Day 15, doubling of blast count % in blood from baseline; death determined to be related to disease or disease progression; and investigator reported disease progression.
Time Frame: Baseline up to 28 days after the last dose, up to approximately 3 years
Population: Disease response was assessed in the Intent-to-Treat Population.
Measure: Count of Participants; unit: Participants
Groups:
- Quizartinib 12 mg ID: Participants received quizartinib (AC220) 12 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 18 mg ID: Participants received quizartinib (AC220) 18 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 27 mg ID: Participants received quizartinib (AC220) 27 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 40 mg ID: Participants received quizartinib (AC220) 40 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 60 mg ID: Participants received quizartinib (AC220) 60 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 90 mg ID: Participants received quizartinib (AC220) 90 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 135 mg ID: Participants received quizartinib (AC220) 135 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 200 mg ID: Participants received quizartinib (AC220) 200 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 300 mg ID: Participants received quizartinib (AC220) 300 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 450 mg ID: Participants received quizartinib (AC220) 450 mg/day on an intermittent dosing (ID) schedule.
- Quizartinib 200 mg CD: Participants received quizartinib (AC220) 200 mg/day on a continuous dosing (CD) schedule.
- Quizartinib 300 mg CD: Participants received quizartinib (AC220) 300 mg/day on a continuous dosing (CD) schedule.
- All Participants: All participants who received quizartinib, regardless of dosage and dosing schedule.
Arm/Group | Quizartinib 12 mg ID | Quizartinib 18 mg ID | Quizartinib 27 mg ID | Quizartinib 40 mg ID | Quizartinib 60 mg ID | Quizartinib 90 mg ID | Quizartinib 135 mg ID | Quizartinib 200 mg ID | Quizartinib 300 mg ID | Quizartinib 450 mg ID | Quizartinib 200 mg CD | Quizartinib 300 mg CD | All Participants
Number analyzed (Participants) | 3 | 8 | 6 | 5 | 5 | 3 | 5 | 6 | 4 | 6 | 17 | 8 | 76
Participants | 2 | 2 | 3 | 3 | 2 | 1 | 1 | 1 | 2 | 2 | 4 | 3 | 26

4. Secondary Outcome: Number of Participants Achieving a Best Disease Response by Dose Cohort in Terms of Best Overall Response Following Oral Administration of Quizartinib in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Complete Response (CR) response criteria included either a post-baseline bone marrow (BM) biopsy or aspiration % blasts <5%, absolute neutrophil count (ANC) >1×10^9/L and platelet count >100×10^9/L on the same date as the qualifying BM assessment. CRp response included all CR criteria met, except participant did not experience a platelet recovery (ANC recovery required). CRi response included a qualifying BM result, but not an ANC recovery. Participants may or may not have had a platelet recovery and were not required to be transfusion independent. Partial remission (PR) response included a decrease of ≥50% in % blasts in the BM aspirate or biopsy from baseline to a post-baseline result between 5% to 25% in the bone marrow aspirate or biopsy. Nonresponders (NR) had a pre- and 1 or more post-baseline BM assessment carried out, but results did not meet any response criteria. Participants who were not evaluable (NE) did not have at least 14 days of treatment and were not assessed.
Time Frame: Baseline up to 28 days after the last dose, up to approximately 3 years
Population: Disease response was assessed in the Intent-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib 12 mg ID | Quizartinib 18 mg ID | Quizartinib 27 mg ID | Quizartinib 40 mg ID | Quizartinib 60 mg ID | Quizartinib 90 mg ID | Quizartinib 135 mg ID | Quizartinib 200 mg ID | Quizartinib 300 mg ID | Quizartinib 450 mg ID | Quizartinib 200 mg CD | Quizartinib 300 mg CD | All Participants
Number analyzed (Participants) | 3 | 8 | 6 | 5 | 5 | 3 | 5 | 6 | 4 | 6 | 17 | 8 | 76
Participants
  Overall response | 0 | 1 | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 6 | 2 | 23
  composite CR (CR+CRp+CRi) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 5 | 1 | 10
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  CR with incomplete platelet recovery | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  CR with incomplete hematologic recovery | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 5
  Partial remission (PR) | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 13
  Nonresponder (NR) | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 2 | 5 | 2 | 19
  Not evaluable (NE) | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 8

5. Secondary Outcome: Number of Participants Achieving a Best Disease Response by Dose Cohort in Terms of Progressive Disease Following Oral Administration of Quizartinib in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: as for outcome 3
Time Frame: Baseline up to 28 days after the last dose, up to approximately 3 years
Population: Disease response was assessed in the Evaluable Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib 12 mg ID | Quizartinib 18 mg ID | Quizartinib 27 mg ID | Quizartinib 40 mg ID | Quizartinib 60 mg ID | Quizartinib 90 mg ID | Quizartinib 135 mg ID | Quizartinib 200 mg ID | Quizartinib 300 mg ID | Quizartinib 450 mg ID | Quizartinib 200 mg CD | Quizartinib 300 mg CD | All Participants
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 5 | 2 | 4 | 5 | 4 | 4 | 12 | 7 | 59
Participants | 2 | 2 | 2 | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 3 | 18

6. Secondary Outcome: Number of Participants Achieving a Best Disease Response by Dose Cohort in Terms of Best Overall Response Following Oral Administration of Quizartinib in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Complete Response (CR) response criteria included either a post-baseline bone marrow biopsy or aspiration % blasts <5%, absolute neutrophil count (ANC) >1×10^9/L and platelet count >100×10^9/L on the same date as the qualifying bone marrow assessment. CRp response included all CR criteria met except participant did not experience a platelet recovery. Participants must have experienced an ANC Recovery. CRi response included a qualifying bone marrow result, but did not experience an ANC recovery. Participants may or may not have experienced a platelet recovery and were not required to be transfusion independent. Partial remission (PR) response included a decrease of ≥50% in % blasts in the bone marrow aspirate or biopsy from baseline to a post-baseline result between 5% to 25% in the bone marrow aspirate or biopsy. Nonresponders (NR) had a pre- and 1 or more post-baseline bone marrow assessment carried out, but results did not meet any of the CR or PR or progressive disease criteria.
Time Frame: Baseline up to 28 days after the last dose, up to approximately 3 years
Population: Disease response was assessed in the Evaluable Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib 12 mg ID | Quizartinib 18 mg ID | Quizartinib 27 mg ID | Quizartinib 40 mg ID | Quizartinib 60 mg ID | Quizartinib 90 mg ID | Quizartinib 135 mg ID | Quizartinib 200 mg ID | Quizartinib 300 mg ID | Quizartinib 450 mg ID | Quizartinib 200 mg CD | Quizartinib 300 mg CD | All Participants
Number analyzed (Participants) | 3 | 5 | 4 | 4 | 5 | 2 | 4 | 5 | 4 | 4 | 12 | 7 | 59
Participants
  Overall response | 0 | 1 | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 6 | 2 | 22
  Composite CR (CR+CRp+CRi) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 5 | 1 | 10
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  CR with incomplete platelet recovery | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  CR with incomplete hematologic recovery | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 5
  Partial remission | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 12
  Nonresponder | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 2 | 5 | 2 | 19

7. Secondary Outcome: Number of Participants With Hematologic Improvement Following Oral Administration of Quizartinib in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Hematologic improvement is summarized in terms of Erythroid Response (HI-E), Platelet Response (HI-P), Neutrophil Response (HI-N), and Hematologic Improvement (HI).
  For post-treatment results, HI-E major responders had >2 g/dL increase in hemoglobin for at least 1 result after first treatment and transfusion independent; minor responders 1 to 2 g/dL increase in hemoglobin for at least 1 result post first treatment and a 50% decrease in red blood cell transfusion requirements. For HI-P, major responders had ≥30 × 10^9/L increase in platelet count and transfusion independent; minor responders had 50% or more increase in platelet count with a net increase between 10 to 30 × 10^9/L and 50% decrease in platelet transfusion requirements. For HI-N, major responders had an increase in absolute neutrophil count (ANC) of 100% or an absolute increase of more than 0.5 × 10^9/L (whichever is greater); minor responders had an increase in ANC of 100% but an absolute increase of <0.5 × 10^9/L.
Time Frame: Baseline up to 28 days after the last dose, up to approximately 3 years
Population: Hematologic improvement was assessed in the Intent-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib
Number analyzed (Participants) | 76
Participants
  Erythroid Response (HI-E) Responders: number analyzed (Participants) | 69
  Erythroid Response (HI-E) Responders | 35
  Erythroid Response (HI-E) Major Responders: number analyzed (Participants) | 69
  Erythroid Response (HI-E) Major Responders | 15
  Erythroid Response (HI-E) Minor Responders: number analyzed (Participants) | 69
  Erythroid Response (HI-E) Minor Responders | 20
  Erythroid Response (HI-E) No Response: number analyzed (Participants) | 69
  Erythroid Response (HI-E) No Response | 34
  HI-E Participants excluded | 7
  Platelet Response (HI-P) Responders: number analyzed (Participants) | 68
  Platelet Response (HI-P) Responders | 39
  Platelet Response (HI-P) Major Responders: number analyzed (Participants) | 68
  Platelet Response (HI-P) Major Responders | 18
  Platelet Response (HI-P) Minor Responders: number analyzed (Participants) | 68
  Platelet Response (HI-P) Minor Responders | 21
  Platelet Response (HI-P) No Response: number analyzed (Participants) | 68
  Platelet Response (HI-P) No Response | 29
  HI-P Participants excluded | 8
  Neutrophil Response (HI-N) Responders: number analyzed (Participants) | 50
  Neutrophil Response (HI-N) Responders | 26
  Neutrophil Response (HI-N) Major Responders: number analyzed (Participants) | 50
  Neutrophil Response (HI-N) Major Responders | 19
  Neutrophil Response (HI-N) Minor Responders: number analyzed (Participants) | 50
  Neutrophil Response (HI-N) Minor Responders | 7
  Neutrophil Response (HI-N) No Response: number analyzed (Participants) | 50
  Neutrophil Response (HI-N) No Response | 24
  HI-N Participants excluded: number analyzed (Participants) | 50
  HI-N Participants excluded | 26
  Hematologic Improvement (HI) Responders: number analyzed (Participants) | 75
  Hematologic Improvement (HI) Responders | 60
  Hematologic Improvement (HI) Any Major Response: number analyzed (Participants) | 75
  Hematologic Improvement (HI) Any Major Response | 38
  Hematologic Improvement (HI) Any Minor Response: number analyzed (Participants) | 75
  Hematologic Improvement (HI) Any Minor Response | 22
  HI Participants excluded | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from after initiation of study drug up to 30 days after last dose, up to approximately 3 years.
Arm/Group | Quizartinib 12 mg ID | Quizartinib 18 mg ID | Quizartinib 27 mg ID | Quizartinib 40 mg ID | Quizartinib 60 mg ID | Quizartinib 90 mg ID | Quizartinib 135 mg ID | Quizartinib 200 mg ID | Quizartinib 300 mg ID | Quizartinib 450 mg ID | Quizartinib 200 mg CD | Quizartinib 300 mg CD
All-Cause Mortality (participants affected / at risk) | 3/3 | 8/8 | 6/6 | 5/5 | 5/5 | 3/3 | 5/5 | 5/6 | 4/4 | 6/6 | 16/17 | 8/8
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/8 | 1/6 | 3/5 | 4/5 | 2/3 | 4/5 | 3/6 | 3/4 | 5/6 | 9/17 | 8/8
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 5/6 | 5/5 | 5/5 | 3/3 | 5/5 | 6/6 | 4/4 | 6/6 | 15/17 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quizartinib 12 mg ID (N=3) | Quizartinib 18 mg ID (N=8) | Quizartinib 27 mg ID (N=6) | Quizartinib 40 mg ID (N=5) | Quizartinib 60 mg ID (N=5) | Quizartinib 90 mg ID (N=3) | Quizartinib 135 mg ID (N=5) | Quizartinib 200 mg ID (N=6) | Quizartinib 300 mg ID (N=4) | Quizartinib 450 mg ID (N=6) | Quizartinib 200 mg CD (N=17) | Quizartinib 300 mg CD (N=8)
Disease progression (General disorders) | 0 | 2 | 0 | 1 | 4 | 1 | 1 | 2 | 1 | 4 | 5 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis fungal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haemtoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quizartinib 12 mg ID (N=3) | Quizartinib 18 mg ID (N=8) | Quizartinib 27 mg ID (N=6) | Quizartinib 40 mg ID (N=5) | Quizartinib 60 mg ID (N=5) | Quizartinib 90 mg ID (N=3) | Quizartinib 135 mg ID (N=5) | Quizartinib 200 mg ID (N=6) | Quizartinib 300 mg ID (N=4) | Quizartinib 450 mg ID (N=6) | Quizartinib 200 mg CD (N=17) | Quizartinib 300 mg CD (N=8)
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 3 | 2 | 2 | 5 | 1 | 4 | 6 | 2
Pyrexia (General disorders) | 0 | 3 | 1 | 3 | 2 | 1 | 1 | 3 | 2 | 1 | 7 | 3
Fatigue (General disorders) | 0 | 0 | 2 | 2 | 2 | 1 | 3 | 3 | 2 | 3 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 3 | 1 | 4 | 4 | 3
Disease progression (General disorders) | 0 | 2 | 0 | 1 | 4 | 1 | 1 | 2 | 1 | 4 | 5 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 2 | 3 | 0 | 1 | 2 | 2 | 2 | 5 | 3
Odema peripheral (General disorders) | 1 | 1 | 2 | 1 | 2 | 2 | 2 | 3 | 2 | 1 | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 3 | 7 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 1 | 3 | 3 | 2 | 0 | 1 | 1 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 4 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 3
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 0 | 2 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 3 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 4 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 0
ECG QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 1
Chills (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No